CLINICAL TRIAL: NCT07360496
Title: Investigation of the Relationships Between Core Endurance, Finger Grip Strength, Fatigue, and Hand Function in Patients With Rheumatoid Arthritis
Brief Title: Core Endurance, Finger Grip Strength, Fatigue, and Hand Function in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Selvin BALKİ, Principal Investigator, Cumhuriyet University
Other Study IDs: SCU-FTR-SB-05
Record Dates: First submitted 2026-01-09; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis; Healthy Control
Keywords: Rheumatoid Arthritis; Core Endurance; Pinchmeter; Grip Strength; Fatigue
MeSH Terms: conditions — Arthritis, Rheumatoid; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RA group: Core endurance, finger grip strength, hand function, fatigue, physical activity level, and disease activity were evaluated in patients diagnosed with RA.
- Healthy controls: Core endurance, finger grip strength, hand function, fatigue, and physical activity level were evaluated in healthy control

INTERVENTIONS:
Other:  — Only measurements were taken.

SUMMARY:
This study investigated the relationships between core endurance, finger grip strength, fatigue, and hand function in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
The aim was to evaluate the level of RA activity and disease activity and to examine the differences between healthy controls and RA patients in terms of these results.

A total of 113 people participated in the study, including 75 patients (57 women and 18 men; mean age: 48.65±12.53) diagnosed with RA (moderate and high levels of disease activity) aged 18-65 years and 38 healthy control group members (28 women and 10 men; mean age: 45.11±10.6).

In the evaluation, finger grip strength measurements (double grip, lateral grip, three-point grip) were done using a pinchmeter. In the kor endurance measurement, the patient was asked to lift their knees off the ground in a crawling position by contracting their kor muscles and keeping their waist at a certain distance, and the time they maintained the position was recorded. Hand function with SACRAH (Skor For Assessment And Quantification Of Chronic Rheumatic Affections Of The Hands), fatigue severity with FSS (Fatigue Severity Skor) and physical activity level with FIT Index (Frequency-Intensity-Time) were measured.

ELIGIBILITY:
* RA Group Inclusion Criteria:

  * Diagnosed with RA according to ACR/EULAR criteria
  * Between 18-65 years of age
  * Willing to participate in the study

RA Group Exclusion Criteria:

* Having any chronic disease other than RA
* Having another musculoskeletal disease
* Having adaptation problems and psychiatric illnesses that would impair participation in the study
* Having hearing loss that would impair communication
* Having severe vision loss
* Having another rheumatic disease other than RA
* Having any uncontrolled cardiopulmonary disease
* Having a serious deformity or severe pain in the extremities or trunk that would prevent taking a crawling position (7 or higher on a 10-point numerical pain scale) (being present)
* Hand deformity or pain severe enough to prevent finger grip strength measurements
* History of any serious trauma or injury within the last 6 months
* Changes in medication used for RA within the last 3 months
* Receiving physiotherapy or other treatment other than medication
* History of musculoskeletal surgery (trunk, extremities)
* Being pregnant or breastfeeding

Health Controls Inclusion Criteria:

* Being between 18-65 years of age
* Voluntary participation in the study Health Controls Exclusion Criteria: ● Having any diagnosed illness
* Having a history of trauma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients RA diagnosis and health Controls
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-09-09 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Core endurance | December 2022-September 2023
  Modified prone plank. This test began with a crawling position, and the participant was instructed to lift their knees off the ground and maintain that position.

SECONDARY OUTCOMES:
Finger grip strength | December 2022-September 2023
  Finger grip strength (double grip, lateral grip, three-point grip) was measured using a pinchmeter.
Hand function | December 2022-September 2023
  Hand function was measured with SACRAH (Score For Assessment And Quantification Of Chronic Rheumatic Affections Of The Hands). SACRAH is a scale consisting of 23 questions. Questions 1-17 assess hand function, questions 18-19 assess stiffness, and questions 20-23 assess pain. Scoring is done on a scale of 0-100, and the higher the score, the worse the outcome.
Fatigue severity | December 2022-September 2023
  Fatigue severity was determined using FSS (Fatigue Severity Score).It contains 9 questions, each scored between 0-7. A total FSS score of 6.1 or higher indicates chronic fatigue.
Physical activity level | December 2022-September 2023
  Determined with FIT Index (Frequency-Intensity-Time).The maximum FIT index score is 100. Higher FIT scores indicate high levels of physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No